CLINICAL TRIAL: NCT06755372
Title: The Role of Toll-like Receptor-4 in Periodontitis Patients With End-stage Renal Disease in a Sample of Egyptian Population
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Other Study IDs: R-625
Record Dates: First submitted 2024-12-31; First posted 2025-01-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis; End-stage Renal Disease
Keywords: Chronic Kidney Disease; End-Stage Renal Disease; Periodontitis; Toll-like Receptor 4; Genetic Polymorphism
MeSH Terms: conditions — Periodontitis; Kidney Failure, Chronic; Renal Insufficiency, Chronic; Macular Degeneration, Age-Related, 10

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood Samples:
  Whole blood collected in EDTA-containing vacutainer tubes. This is essential for extracting genomic DNA.
  DNA Samples:
  Genomic DNA extracted from the collected blood samples. These DNA samples will be used for genetic analysis, including SNP genotyping in the TLR4 gene.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Subjects with Periodontitis: Description: This group consists of 50 systemically healthy individuals diagnosed with periodontitis. Participants are of both genders, aged between 30 and 60 years. They have Periodontitis stage II and/or stage III and do not have any history of systemic diseases or long-term medication use. All smokers were excluded from this group.
  Interventions of Interest:
  Clinical assessment of periodontal parameters such as Plaque Index (PI), Gingival Index (GI), Probing Depth (PD), and Clinical Attachment Level (CAL) using standard methods.
  Evaluation of the proportion of bleeding sites as a Bleeding on Probing (BOP) score.
- ESRD Patients with Periodontitis: Description: This group includes 50 individuals diagnosed with end-stage renal disease (ESRD) who are on regular hemodialysis. Participants are of both genders, aged between 30 and 60 years, and unrelated Egyptians from similar socioeconomic statuses residing in the same geographical area. They also suffer from Periodontitis stage II and/or stage III. All participants have underlying type 2 diabetes mellitus. Exclusions include those with kidney transplants, other systemic diseases except diabetes, history of malignancy, and smokers.
  Interventions of Interest:
  Clinical assessment of periodontal parameters similar to Group I, including PI, GI, PD, and CAL.
  Analysis of genetic variations in the TLR4 gene through blood sample collection and DNA extraction.
  SNP genotyping in the TLR4 gene performed using Real Time Polymerase Chain Reaction (RT-PCR).

SUMMARY:
Chronic kidney disease (CKD) is a significant public health issue in Egypt, leading to end-stage renal disease (ESRD). ESRD patients often suffer from oral abnormalities due to the disease and medications. Periodontitis is linked to systemic diseases, including renal disease, with inflammation playing a key role. TLR4 genetic variations may influence susceptibility to CKD and periodontitis. This study investigates the association between TLR4 [Gly/Thr (rs2149356)] polymorphism and chronic periodontal disease in ESRD patients in Egypt.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD), which ranks sixth among the top causes of death from 2009 to 2019, has become 36% more prevalent in Egypt, following the global trend (The Center for Economic and Social Rights: 2021).

Since untreated CKD can lead to end-stage renal disease (ESRD), which is the complete loss of renal function when patients are dialysis-dependent and require a kidney transplant, CKD has emerged as a significant public health issue in Egypt (Chen et al., 2024).

According to the most recent data available, the prevalence of dialysis in Egypt was 0.61 per 1000 persons in 2019; the incidence was estimated to be 0.19 per 1000 people (Bello et al., 2029; Farag et al., 2022).

ESRD patients exhibit a variety of oral abnormalities, as the disease and the medications taken by those patients might exacerbate or cause the development of caries, periodontal disease, mucosal lesions, decreased saliva production, and other oral disorders (Trzcionka et al., 2020).

Periodontitis is a widely prevalent inflammatory and infectious disease affecting the supporting structure of the teeth. In the past few decades, the association between periodontitis and systemic diseases has received much attention (Abou-Bakr et al., 2022; Mainas et al., 2022).

There is increasing evidence to suggest that renal disease and periodontitis are strongly correlated (Kapellas et al., 2019; Li et al., 2021). Furthermore, periodontitis has been implicated in the decline in renal function, cardiovascular outcomes, and also mortality of CKD patients (Lertpimonchai et al., 2019; Tai et al., 2021).

Apart from inadequate oral hygiene and the prevalence of inflammatory diseases, renal osteodystrophy, elevated urea levels, alterations in salivary composition, and host factors linked to underlying systemic diseases that modify the host's reaction to periodontal infection are additional factors that accelerate periodontal disease in patients with ESRD (Pakpour et al., 2015).

While CKD susceptibility is known to be influenced by traditional risk factors, such as age, hypertension, diabetes, and dyslipidemia, emerging evidence indicates that nontraditional risk factors, such as chronic inflammation-mediated activation of the innate immune system, also contribute to the pathogenesis of CKD and diabetic nephropathy (DN) (Lin and Tang, 2014; Verzola et al., 2014).

Toll-like receptor 4 (TLR4) is one of the key components of the mammalian innate immune system. Binding of exogenous and endogenous ligands activates TLR4, which in turn triggers a signaling cascade, leading to initiation of an adaptive and innate immune response. Genetic variations in TLR4 are thought to alter the ligand-binding capacity and contribute to the chronic inflammation-mediated pathogenesis of many diseases (Noreen and Arshad, 2015).

TLR4 binds to the exogenous ligands, such as hyaluronan, heparan sulfate, or fibrinogen, and promotes renal injury by increasing inflammation (Lin and Tang, 2014). Chronic inflammation-mediated activation of the innate immune system has been implicated in the pathogenesis of CKD/DN. In diabetes, TLR4 may sense high glucose, free fatty acids, and advanced glycation end products as signal molecules and trigger the inflammatory signaling cascade to contribute to DN (Verzola et al., 2014).

In DN patients, TLR4 expression was found to be upregulated in glomeruli with a subsequent decline in eGFR. TLR4 expression was associated with increased expression of TGF-β1 in kidney biopsies from patients with CKD/DN (Lepenies et al., 2011). In summary, it is evident that TLR4 activation likely contributes to DN (Thameem et al., 2016).

According to Murphy et al. (1993), genetic predisposition is the difference in immune-related DNA molecules within the host that influences the development and occurrence of disease. Investigating the variations in immune-related molecules responsible for susceptibility and prevention of periodontitis is crucial because a set of host genetic variants may contribute to the occurrence and development of chronic periodontitis by selectively engaging in the pathophysiological process (Gordon et al., 2002).

Immunologically competent cells express a class of trans membrane proteins known as Toll-like Receptors (TLRs) (Medzhitov et al., 1997). They identify and bind MAMPs, or microorganism-associated molecular patterns, which are produced by bacteria and are important molecules for the eradication of microbes (Takeda et al., 2003).

TLR4 is also expressed in gingival epithelial keratinocytes, fibroblasts, and antigen-presenting cells. Lipopolysaccharide (LPS) of Gram-negative bacteria periopathogens, such as Porphyromonas gingivalis, Aggregatibacter actinomycetemcomitans, and Veillonella parvula, has been demonstrated to be specifically recognized by TLR4. These bacteria collaborate with multiple protein components, including lipopolysaccharide binding protein (LBP) and CD14 (Yoshimora et al., 2002; Mori et al., 2003).

According to Uematsu S. et al. (2008), this causes the NF-kB pathway to activate the inflammatory cells, which in turn activates the cytokine network. Bone loss symptoms are caused by cytokines such IL-6, IL-8, and TNF-α, as well as matrix metalloproteinase and prostaglandin E2. (Giannobile et al., 2008). Additionally, in a periodontal paradigm, TLR-4-deficient C3H/HeJ mice showed decreased bone resorption, suggesting that TLRs may be essential for the development and susceptibility of periodontitis (Hou et al., 2009).

The TLR4 genes' single nucleotide polymorphisms (SNPs) have been shown to result in reduced cytokine production by epithelial cells in response to LPS stimulation and impaired microbe detection (Schroder et al., 2005). Hence, after being stimulated by bacteria in periodontal tissues, TLRs take part in innate immune responses and inflammatory reactions. Nonetheless, there is disagreement on the degree to which these receptors influence individual variations in periodontitis susceptibility (Ding et al., 2015).

Through a variety of pattern-recognition receptors, the host immune system predominantly identifies invasive infections. These receptors identify pathogen-associated molecular patterns (PAMPs) that are conserved and generally shared by broad assemblages of microorganisms, such as lipopolysaccharide-producing bacteria (Folwaczny et al., 2004).

The transmembrane receptors known as Toll-like receptors belong to the evolutionary conserved interleukin-1 super-family and are capable of identifying molecular patterns linked to pathogens (Takeda K, Akira, 2003). The Toll/IL-1R (TIR) domain refers to the cytoplasmic domain of Toll-like receptors that exhibits strong similarities to the intracellular region of the interleukin-1 (IL-1) receptor family (Aderem and Ulevitch, 2000).

Leucine-rich repeats (LRRs) are present in the Toll-like receptor extracellular domain.Lipopolysaccharide is the primary cause of inflammation in gram-negative bacterial infections, and Toll-like receptor-4 plays a critical role in mediating its effects, which include activating the inflammatory molecular cascade through the NFκB pathway (Medzhitov et al., 1997). Lipopolysaccharide-binding protein (LBP), the CD14 receptor, and the MD-2 protein are three additional molecules that are necessary for the identification and transmission of the lipopolysaccharide signal through the Toll-like receptor-4. Numerous other organs, including endothelial cells, macrophages, cardiomyocytes, and airway epithelia, express the TLR-4 protein. (Zarember and Godowski 2002).

Two frequently occurring segregating missense variants that impact the extracellular domain of the TLR4 protein have been identified: Asp299Gly and Thr399Ile (Arbour et al., 2000). The two mutations cause LPS signaling to be less effective and less able to cause inflammation. Individuals with these mutations were consistently found to have an elevated risk of gram-negative infections and a much lower risk of atherosclerosis. (Agnese et al., 2002).

Since TLR4 is a crucial mediator between pathogen-produced substances and the start of host defense, variations in the TLR4 gene may play a significant role in an individual's vulnerability to bacterial infections, which in turn may have an impact on the inflammatory process (Akira et al., 2003).

TLR4 SNPs have also been demonstrated to affect the risk of various multifactorial disorders. These findings suggest that TLR4 gene sequence variants with abnormal function, may contribute to the development of various diseases, including multifactorial disorders (Shibuya et al., 2008).

In a previous study by Farouk et al., 2021, it was concluded that TLR4 SNP rs2149356 was linked with chronic periodontitis in an Egyptian sample. Thus, the aim of the present study is to investigate the association between the genetic variations of TLR-4 [Gly/Thr (rs2149356)] and chronic periodontal disease in ESRD. To the best of the authors knowledge, no published studies from the Middle East and North Africa region exist, and there's a gap of knowledge in the role of the TLR-4 [Gly/Thr (rs2149356)] gene polymorphism in relation to ESRD patients with chronic periodontitis in the North African Egyptian subjects.

ELIGIBILITY:
Group I: Healthy Subjects with Periodontitis

Inclusion Criteria:

Age: 30 to 60 years

Gender: Both male and female

Diagnosed with Periodontitis stage II and/or stage III

Systemically healthy, no history of systemic diseases

Not on long-term medications

Exclusion Criteria:

Smokers

Individuals with any systemic disease or long-term medication use

Group II: ESRD Patients with Periodontitis

Inclusion Criteria:

Age: 30 to 60 years

Gender: Both male and female

Diagnosed with end-stage renal disease (ESRD) on regular hemodialysis

Diagnosed with Periodontitis stage II and/or stage III

Unrelated Egyptians from a similar socioeconomic status, residing in the same geographical area

Underlying type 2 diabetes mellitus

Exclusion Criteria:

Individuals with kidney transplants

Individuals with systemic diseases other than diabetes

History of malignancy

Smokers

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group I: Healthy Subjects with Periodontitis Number of Participants: 50 These individuals were systemically healthy but had periodontal disease. They were recruited from the Periodontology Clinic at the Faculty of Dentistry, Fayoum University.
  Group II: ESRD Patients with Periodontitis Number of Participants: 50 Description: These individuals had ESRD and periodontal disease. They were recruited from the hemodialysis center at Benha University Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL): | single point "Baseline"
  Description: The CAL measures the extent of periodontal support around a tooth, from the cementoenamel junction (CEJ) to the base of the pocket, crucial for diagnosing periodontal disease.
  Measurement Method: CAL is recorded using a periodontal probe by measuring probing depth (PD) and distance from the gingival margin to the CEJ. CAL is calculated as follows:
  CEJ at gingival margin: CAL = PD Gingival margin coronal to CEJ: CAL = PD - Distance from Gingival Margin to CEJ Gingival margin apical to CEJ: CAL = PD + Distance from CEJ to Gingival Margin in non- periodontitis individuals CAL is zero

SECONDARY OUTCOMES:
Bleeding on Probing (BOP) | single point "Baseline"
  Description: BOP is a clinical measurement used to assess gingival inflammation. It indicates the presence of bleeding in the gums after they are gently probed, reflecting the health of the gingival tissues.
  Measurement Method: A standardized manual probe with controlled force is used to probe the bottom of the sulcus or periodontal pocket at six locations around each tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual). The presence or absence of bleeding is recorded within 10 seconds of probing.

OTHER OUTCOMES:
Genetic Analysis - TLR4 SNP Genotyping | single point "Baseline"
  Description: This analysis involves genotyping single nucleotide polymorphisms (SNPs) in the TLR4 gene, which plays a crucial role in the immune response by recognizing pathogen-associated molecular patterns.
  Measurement Method: DNA is extracted from blood samples, and specific SNPs in the TLR4 gene (e.g., rs2149356, Asp299Gly rs4986790, and Thr399Ile rs4986791) are analyzed using Real-Time Polymerase Chain Reaction (RT-PCR). This helps determine the genetic variations associated with periodontal disease in patients.
  kits might have a detection range from 0.156 ng/mL to 10 ng/mL for TLR4 protein detection

CONTACTS AND LOCATIONS:
Overall Officials: Fatma E. A. Hassanein, PHD, Principal Investigator — king Salman Intwenational University University
Locations (1):
- hemodialysis center at Benha University Hospital., Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided